CLINICAL TRIAL: NCT01273181
Title: Phase I/II Study of Metastatic Cancer That Expresses MAGE-A3/12 Using Lymphodepleting Conditioning Followed by Infusion of Anti-MAGE-A3/12 TCR-Gene Engineered Lymphocytes
Brief Title: MAGE-A3/12 Metastatic Cancer Treatment With Anti-MAGE-A3/12 TCR-Gene Engineered Lymphocytes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110062; 11-C-0062
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Cancer; Metastatic Renal Cancer; Metastatic Melanoma
Keywords: Immunotherapy; Gene Therapy; Metastatic Cancer; Clinical Response; Metastatic Melanoma; Metastatic Renal Cell Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — aldesleukin; Interleukin-2; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ph I:Anti-MAGE A3/12 TCR PBL 5x10e9 (Experimental): Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Note for phase I: The study will begin by evaluating the safety of two ranges of cells, 5x10^9-3x10^10, and greater than 3x10^10-1x10^11 in a standard phase I dose escalation fashion using a 3+3 design.
  Interventions: Biological: PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes; Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine
- Ph I:Anti-MAGE A3/12 TCR PBL 3x10e10 (Experimental): Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Note for phase I: The study will begin by evaluating the safety of two ranges of cells, 5x10^9-3x10^10, and greater than 3x10^10-1x10^11 in a standard phase I dose escalation fashion using a 3+3 design.
  Interventions: Biological: PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes; Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine
- Ph II:Anti-MAGE TCR PBL MTD+HD IL-2 (Experimental): Phase II:Anti-MAGE A3/12 TCR PBL MTD + HD IL-2, Melanoma, RCC
  Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Note for phase II:patients will be entered into two cohorts based on histology:cohort 1 will include patients with metastatic melanoma or renal cell cancer; cohort 2 will include patients with other types of metastatic cancer.
  Interventions: Biological: PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes; Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine
- Ph II:Anti-MAGE A3/12 TCR PBL MTD (Experimental): Phase II: Anti-MAGE A3/12 TCR PBL MTD + HD-IL2 Other Cancer
  Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Note for phase II:patients will be entered into two cohorts based on histology:cohort 1 will include patients with metastatic melanoma or renal cell cancer; cohort 2 will include patients with other types of metastatic cancer.
  Interventions: Biological: PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes; Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes
Drug: Aldesleukin — 720,000 IU/kg every 8 hours for a maximum of 15 doses
  Other Names: IL-2
Drug: Cyclophosphamide — 60 mg/kg/day x 2 days intravenous (IV)over 1 hour.
Drug: Fludarabine — 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.

SUMMARY:
Background:

- MAGE-A3/12 is a type of protein commonly found on certain types of cancer cells, particularly in metastatic cancer. Researchers have developed a process to take lymphocytes (white blood cells) from cancer patients, modify them in the laboratory to target cancer cells that contain MAGE-A3/12, and return them to the patient to help attack and kill the cancer cells. These modified white blood cells are an experimental treatment, but researchers are interested in determining their safety and effectiveness as a possible treatment for cancers that involve MAGE-A3/12.

Objectives:

- To evaluate the safety and effectiveness of anti-MAGE-A3/12 lymphocytes as a treatment for metastatic cancers that have not responded to standard treatment.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with metastatic melanoma, renal cell cancer, or another type of metastatic cancer that has not responded to standard treatment.

Design:

* Participants will be screened with a full medical history and physical examination, as well as blood and urine tests, tumor samples, and imaging studies.
* Participants will have leukapheresis to collect enough white blood cells for modification in the laboratory.
* Seven days before the start of anti-MAGE-A3/12 treatment, participants will have chemotherapy with cyclophosphamide and fludarabine to suppress the immune system in preparation for the treatment.
* After the last dose of chemotherapy, participants will receive the anti-MAGE-A3/12 cells as an infusion for 20 to 30 minutes, followed by a dose of interleukin-2 to keep the anti-MAGE-A3/12 cells alive and active as long as possible. Participants will also receive filgrastim to encourage the production of blood cells.
* Participants will remain in the hospital to be monitored for possible side effects, and after release from the hospital will have regular followup exams with blood samples and imaging studies to evaluate the effectiveness of the treatment....

DETAILED DESCRIPTION:
Background

We have constructed a single retroviral vector that contains both alpha and beta chains of a T cell receptor (TCR) that recognizes the MAGE-A3/12 tumor antigen, which can be used to mediate genetic transfer of this TCR with high efficiency (> 30%) without the need to perform any selection.

In co-cultures with human leukocyte antigen serotype within HLA-A serotype group (HLA-A2) and MAGE-A3/12 double positive tumors, anti-MAGE-A3/12 TCR transduced T cells secreted significant amounts of Interferon (IFN)-gamma with high specificity.

Objectives:

Primary objectives:

* Determine if the administration of anti-MAGE-A3/12 engineered peripheral blood lymphocytes and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer that expresses the MAGE-A3/12 antigen.
* Determine the toxicity profile of this treatment regimen

Secondary objectives:

-Determine the in vivo survival of TCR gene-engineered cells.

Eligibility:

Patients who are human leukocyte antigen (HLA)-A*0201 positive and 18 years of age or older must have:

* metastatic cancer whose tumors express the MAGE-A3/12 antigen;
* previously received and have been a non-responder to or recurred following standard care for metastatic disease;

Patients may not have:

-contraindications for high dose aldesleukin administration.

Design:

PBMC obtained by leukapheresis (approximately 10^10) cells) will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.

Transduction is initiated by exposure of approximately 10^7 to 5 X 10^8 cells to retroviral vector supernatant containing the anti-MAGE-A3/12 TCR genes.

The study will begin by evaluating the safety of two ranges of cells, 5 x 10^9 - 3 x 10^10, and greater than 3 x 10^10- 1 x 10^11 in a standard phase I dose escalation fashion using a 3+3 design. Once this safety has been confirmed, patients will be enrolled into the phase 2 portion of the trial using up to 1 x 10^11 cells. In the phase 2 portion, patients will be entered into two cohorts based on histology: cohort 1 will include patients with metastatic melanoma or renal cell cancer; cohort 2 will include patients with other types of metastatic cancer.

Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, TCR gene-transduced peripheral blood mononuclear cells (PBMC) plus intravenous (IV) aldesleukin (720,000 IU/kg every (q)8h for a maximum of 15 doses).

Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment. If the patient has stable disease (SD) or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will continue to be followed with this evaluation every 3-4 months until off study criteria are met.

For each of the 2 strata evaluated in the phase 2 portion, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.

For both strata, the objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-MAGE-A3/12 TCR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% partial response (PR) + complete response (CR) rate (p1=0.20).

ELIGIBILITY:
* INCLUSION CRITERIA:

Metastatic cancer that expresses MAGE-A3/12 as assessed by one of the following methods: reverse transcription polymerase chain reaction (RT-PCR) on tumor tissue defined as 30,000 copies of MAGE-A3/12 per 106 GAPDH copies, or by immunohistochemistry of resected tissue defined as 10% or greater of cells being 2-3+, or serum antibody reactive with MAGE-A3/12. Metastatic cancer diagnosis will be confirmed by the Laboratory of Pathology at the National Cancer Institute (NCI).

Patients with melanoma or renal cell cancer must have previously received high dose aldesleukin and have been either non-responders (progressive disease) or have recurred. Patients with other histologies, must have previously received at least one systemic standard care (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.

Greater than or equal to 18 years of age.

Willing to sign a durable power of attorney

Able to understand and sign the Informed Consent Document

Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.

Life expectancy of greater than three months.

Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.

Patients must be human leukocyte antigen (HLA)-A*0201 positive

Serology:

* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.

Hematology:

* Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
* White blood cell (WBC) (> 3000/mm^3).
* Platelet count greater than 100,000/mm^3.
* Hemoglobin greater than 8.0 g/dl.

Chemistry:

* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
* Serum creatinine less than or equal to 1.6 mg/dl.
* Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

EXCLUSION CRITERIA:

Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.

Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.

Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).

Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).

Concurrent Systemic steroid therapy

History of severe immediate hypersensitivity reaction to any of the agents used in this study.

History of coronary revascularization or ischemic symptoms

Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.

Documented LVEF of less than or equal to 45% tested in patients with:

* History of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
* Age greater than or equal to 60 years old

Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

* A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
* Symptoms of respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenberg SA. Progress in human tumour immunology and immunotherapy. Nature. 2001 May 17;411(6835):380-4. doi: 10.1038/35077246. PMID 11357146
- [Background] Berendt MJ, North RJ. T-cell-mediated suppression of anti-tumor immunity. An explanation for progressive growth of an immunogenic tumor. J Exp Med. 1980 Jan 1;151(1):69-80. doi: 10.1084/jem.151.1.69. PMID 6444236
- [Background] Gattinoni L, Powell DJ Jr, Rosenberg SA, Restifo NP. Adoptive immunotherapy for cancer: building on success. Nat Rev Immunol. 2006 May;6(5):383-93. doi: 10.1038/nri1842. PMID 16622476
- [Derived] Abate-Daga D, Hanada K, Davis JL, Yang JC, Rosenberg SA, Morgan RA. Expression profiling of TCR-engineered T cells demonstrates overexpression of multiple inhibitory receptors in persisting lymphocytes. Blood. 2013 Aug 22;122(8):1399-410. doi: 10.1182/blood-2013-04-495531. Epub 2013 Jul 16. PMID 23861247
- [Derived] Morgan RA, Chinnasamy N, Abate-Daga D, Gros A, Robbins PF, Zheng Z, Dudley ME, Feldman SA, Yang JC, Sherry RM, Phan GQ, Hughes MS, Kammula US, Miller AD, Hessman CJ, Stewart AA, Restifo NP, Quezado MM, Alimchandani M, Rosenberg AZ, Nath A, Wang T, Bielekova B, Wuest SC, Akula N, McMahon FJ, Wilde S, Mosetter B, Schendel DJ, Laurencot CM, Rosenberg SA. Cancer regression and neurological toxicity following anti-MAGE-A3 TCR gene therapy. J Immunother. 2013 Feb;36(2):133-51. doi: 10.1097/CJI.0b013e3182829903. PMID 23377668
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0062.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ph I:study will begin by evaluating the safety of 2 ranges of cells,5x10^9-3x10^10, & >3x10^10-1x10^11 in a standard ph I dose escalation using a 3+3 design. Ph II:pts will be entered into 2 cohorts based on histology:cohort 1 will include pts with metastatic melanoma or RCC; cohort 2 will include pts with other types of metastatic cancer.
Groups:
- Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9; Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10: Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
- Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC: anti-MAGE A3/12 TCR PBL MTD + HD IL-2 Melanoma, RCC
- Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer: anti-MAGE A3/12 TCR PBL MTD + HD IL-2 Other cancers
Period: Phase I, Dose 1
Arm/Group | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer
Started | 3 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Study termination | 1 | 0 | 0 | 0
Period: Phase I, Dose 2
Arm/Group | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer
Started | 0 | 3 | 0 | 0
Completed | 0 | 2 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Death during treatment | 0 | 1 | 0 | 0
Period: Phase 2, Dose 1
Arm/Group | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer
Started | 0 | 0 | 2 | 0
Completed | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Study termination | 0 | 0 | 1 | 0
Period: Phase 2, Dose 2
Arm/Group | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer
Started | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1
Not completed — Death during treatment | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC: Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC
  Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
- Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer: Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer
  Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
- Total: Total of all reporting groups
Arm/Group | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer | Total
Number analyzed (Participants) | 3 | 3 | 2 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 0 | 8
  >=65 years | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (11.4) | 39.7 (16.9) | 62.0 (0.0) | 71.0 | 51.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 5
  Male | 1 | 2 | 1 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 2 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 00 | 0 | 0 | 0
  White | 3 | 3 | 2 | 1 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Toxicity Profile
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer
Number analyzed (Participants) | 3 | 3 | 2 | 1
Participants | 3 | 3 | 2 | 1

2. Primary Outcome: Clinical Tumor Regression (Complete Response (CR) + Partial Response (PR)) in Patients With Metastatic Cancer
Description: Tumor regression response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is a disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: 2 years
Measure: Number; unit: Participants
Groups:
- Anti-MAGE TCR PBL 5x10e9 +HD IL-2: anti-MAGE A3/12 TCR PBL 3x10e10 to 1 x 10e11 + HD IL-2
  Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
- Anti-MAGE TCR PBL 5x10e10 +HD IL-2: anti-MAGE A3/12 TCR PBL 5x10e9 to 3 x 10e10 + HD IL-2
  Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
- Anti-MAGE TCR PBL+HD IL-2, Mel, RCC: anti-MAGE A3/12 TCR PBL MTD + HD IL-2 Melanoma, RCC
  Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
- Anti-MAGE TCR PBL +HD IL-2, Other: anti-MAGE A3/12 TCR PBL MTD +HD-IL-1 Other cancers
  Cyclophosphamide : 60 mg/kg/day x 2 days intravenous (IV)
  Aldesleukin : 720,000 IU/kg every 8 hours for a maximum of 15 doses
  PG13-MAGE-A3 TCR9W11 (anti-MAGE-A3/12 TCR) Transduced Autologous Peripheral Blood Lymphocytes :
  Fludarabine : 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
Arm/Group | Anti-MAGE TCR PBL 5x10e9 +HD IL-2 | Anti-MAGE TCR PBL 5x10e10 +HD IL-2 | Anti-MAGE TCR PBL+HD IL-2, Mel, RCC | Anti-MAGE TCR PBL +HD IL-2, Other
Number analyzed (Participants) | 3 | 3 | 2 | 1
Participants
  Complete Response | 1 | 0 | 0 | 0
  Partial Response | 1 | 2 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 (N=3) | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 (N=3) | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC (N=2) | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer (N=1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALT/SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
AST/SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death not associated with CTCAE term (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Speech impairment (e.g. dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Anti-MAGE A3/12 TCR PBL 5x10e9 (N=3) | Phase I:Anti-MAGE A3/12 TCR PBL 3x10e10 (N=3) | Phase II:Anti-MAGE A3/12 TCR PBL MTD+HD IL-2, Melanoma, RCC (N=2) | Phase II: Anti-MAGE A3/12 TCR PBL MTD +HD IL-2, Other Cancer (N=1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 0 (0) — fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular & nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PTT (partial thromboplastin time) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No